CLINICAL TRIAL: NCT01450839
Title: E2022 Patch Formulation Multiple Dose Phase I Study
Brief Title: E2022 Patch Formulation Multiple Dose Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eisai Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Eisai Inc. (Industry)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: E2022-J081-002
Record Dates: First submitted 2011-10-04; First posted 2011-10-12 (Estimated); Last update posted 2012-06-01 (Estimated); Status verified 2012-05

CONDITIONS: Healthy
Keywords: Transdermal Administration; Japanese; elderly; male; volunteers

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (2):
- E2020 5 mg tablet and tape (Experimental)
  Interventions: Drug: E2022
- 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: E2022 — The treatment period consists of 2 periods, Period I and Period II. In Period I, one 5 mg E2020 tablet will be administered in a single dose. In Period II, the tape containing 16 mg E2022 (which corresponds to one 5 mg E2020 tablet) will be applied repeatedly for 17 days. A washout period of at least 8 days will be allowed between the day of single dose administration in Period I and the first day of repeated application in Period II. A post-treatment examination will be performed at least 21 days after the last removal of the investigational product in Period II.
  Arms: E2020 5 mg tablet and tape
Drug: Placebo — Matching Placebo tablets and tape
  Arms: 2

SUMMARY:
This study is to evaluate the safety and tolerability of a E2022 16 mg tape when applied repeatedly for 17 days to healthy elderly Japanese male subjects, using E2022 placebo tape as the control.

ELIGIBILITY:
Inclusion Criteria

1. Subjects who are non-smoking males (not smoking for at least 4 weeks before the administration of the investigational product in Period I) 65 years or older at the time of giving informed consent
2. Subjects whose body mass index (BMI) is 18.5 kg/m^2 to less than 28.0 kg/m^2 at the screening
3. Subjects who give voluntary written consent to participate in the study
4. Subjects who have been fully informed of matters subjects are required to observe during the study and can, and are willing to, comply with the rules.

Exclusion Criteria

1. Subjects with a history of treatment-requiring disease within 8 weeks before administration of the investigational product in Period I or history of infection within 4 weeks before administration of the investigational product in Period I
2. Subjects who have, within 4 weeks before administration of the investigational product in Period I, a disease that might affect the evaluation of the investigational product, such as mental, gastrointestinal, hepatic, renal, respiratory, endocrine, hematological, nervous, or cardiovascular diseases, and inborn error of metabolism
3. Subjects with a history of surgical treatment of the gastrointestinal tract (e.g., resection of the liver, kidney, gastrointestinal tract, etc.) that may affect the pharmacokinetics of the investigational product
4. Subjects with a history of treatment-requiring drug or food allergy or with seasonal allergy at the screening
5. Subjects with a change in body weight of more than 10% at 1 day before investigational product administration in Period I, compared with that observed at the screening
6. Subjects with clinically significant, treatment-requiring symptoms or impairment of organ function, judging from the subjective symptoms/objective findings, vital signs, 12-lead ECG, or laboratory test performed during the period from the screening to immediately before investigational product administration in Period I
7. Subjects with QTc>450 ms on 12-lead ECG performed at the screening or immediately before investigational product administration in Period I
8. Subjects who are positive for human immunodeficiency virus (HIV) antibody, hepatitis B virus surface antigen (HBs antigen), hepatitis C virus (HCV) antibody, or qualitative syphilis test, at the screening
9. Subjects with a history of, or suspected diagnosis of, drug or alcohol dependence or Subjects who are positive for urine drug test at the screening or 1 day before investigational product administration in Period I
10. Subjects who took caffeine-containing or alcoholic beverage within 72 hours before investigational product administration in Period I
11. Subjects who took, within 2 weeks before investigational product administration in Period I, nutritional supplements, herb-containing drug preparations (including Chinese medicines) or other foods or beverages (e.g., grapefruit-containing foods or beverages) that may affect drug-metabolizing enzymes or transporters
12. Subjects who took drug preparations containing St. John's wort within 4 weeks before investigational product administration in Period I
13. Subjects who took prescription drugs within 4 weeks before investigational product administration in Period I
14. Subjects who took non-prescription drugs within 2 weeks before investigational product administration in Period I
15. Subjects who participated in another clinical study within 16 weeks before investigational product administration in Period I and used an investigational product or medical device
16. Subjects who received blood transfusion within 12 weeks, had 400 mL or more whole blood collected within 12 weeks, had 200 mL or more whole blood collected within 4 weeks, or donated blood components within 2 weeks, before investigational product administration in Period I
17. Subjects who performed strenuous exercise at a frequency of 5 days or more per week or who performed, even once, a strenuous exercise lasting 1 hour or more, within 2 weeks before admission for Period I
18. Subjects with past or current clinical signs of cutaneous hypersensitivity or atopic dermatitis to external medicines
19. Subjects in whom the investigational product and the fixing sheet cannot be applied to 6 or more non-overlapping sites on the back (except the vertebral region and the site around the angulus inferior scapulae) by rotation method
20. Subjects with excessive hair at the application site (back)
21. Subjects with conditions at the application site (back), such as skin diseases (e.g., eczema, dermatitis and pigmentary abnormality), external injuries, and scars, that may affect the evaluation of skin symptom
22. Subjects who, or whose partners, are not willing to take reliable contraceptive measures until the completion of the post-treatment examination
23. Subjects who are judged by the investigator or subinvestigator to be inappropriate as subjects of the study

Min Age: 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 16 (Actual)
Dates: Start 2011-09; Primary Completion 2011-11 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Composite (or Profile) of Pharmacokinetics | predose, 0,1, 2, 3, 4, 6, 8,1 2, 24, 48, 72, 96 hours post-dose
  Cmax, Area Under Curve, Tmax

CONTACTS AND LOCATIONS:
Overall Officials: Hidetaka Hiramatsu, Study Director — Neuroscience Cliical Development Section, Japan /Asia Clinical Research PCU
Locations (1):
- Kagoshima, Kagoshima-ken, Japan